CLINICAL TRIAL: NCT00520234
Title: A Randomized, Double-blind, Placebo Controlled Trial of Caspofungin Prophylaxis Followed by Pre-emptive Therapy for Invasive Candidiasis in High-risk Adults in the Critical Care Setting
Brief Title: Randomized Study of Caspofungin Prophylaxis Followed by Pre-emptive Therapy for Invasive Candidiasis in the Intensive Care Unit (ICU)
Acronym: MSG-01
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mycoses Study Group (Network)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Merck, Merck
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MSG-01
Record Dates: First submitted 2007-08-21; First posted 2007-08-23 (Estimated); Results first posted 2011-05-09 (Estimated); Last update posted 2011-05-09 (Estimated); Status verified 2011-04

CONDITIONS: Invasive Candidiasis
Keywords: Candida; Prophylaxis; High risk adults; Intensive care unit (ICU)
MeSH Terms: conditions — Candidiasis, Invasive; Torulopsis | interventions — Caspofungin; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 prophylaxis (Active Comparator): Caspofungin 50 mg Intravenous (IV) daily up to 28 days of therapy
  Interventions: Drug: Caspofungin
- 2 placebo (Placebo Comparator): Normal Saline 100 cc IV daily
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Caspofungin — 50 mg IV daily
  Arms: 1 prophylaxis
Drug: Normal Saline — 100 cc IV daily
  Other Names: placebo
  Arms: 2 placebo

SUMMARY:
Adults admitted to intensive care units are at risk for a variety of complications. Infections due to the fungus called candida are of particular concern. The study will test the possibility that caspofungin, a new therapy for fungal infections, can successfully reduce the rate of candida infections in subjects at risk. It will also test if caspofungin is useful in treating subjects for this disease when diagnosed using a new blood test that is performed twice weekly, permitting earlier diagnosis than current practice standards.

ELIGIBILITY:
Inclusion Criteria:

* Non-pregnant >18 yrs of age
* Subjects admitted to ICU during the preceding 3 days and expected to stay in the ICU for at least another 48 hours.Subjects can be enrolled on days 3-5 of ICU admission.
* Subjects meeting the clinical prediction rule

Exclusion Criteria:

* Subjects with an allergy/intolerance to caspofungin or echinocandin analog
* absolute neutrophil count <500/mm3 at study entry or likely to develop such a count during therapy
* acquired immunodeficiency syndrome, aplastic anemia or chronic granulomatous disease
* moderate or severe hepatic insufficiency
* subjects who are pregnant or lactating
* unlikely to survive < 24 hours
* subjects who have received systemic antifungal therapy within 10 days prior to study entry
* Documented active proven or probable invasive fungal infection upon enrollment
* previously enrolled in this study
* Currently on another investigational agent or have received an investigational agent within 10 days prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2007-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Luis Ostrosky-Zeichner, MD, Principal Investigator — The University of Texas Health Science Center, Houston; Peter G Pappas, MD, Principal Investigator — Mycoses Study Group
Locations (12):
- United States (12):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Southern California, Los Angeles, California
  - University of Colorado, Denver, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Tulane University, New Orleans, Louisiana
  - Harper University Hospital/ Wayne State, Detroit, Michigan
  - Henry Ford Hospital, Detroit, Michigan
  - St. Patrick's Hospital, Missoula, Montana
  - Cooper University Hospital, Camden, New Jersey
  - The Ohio State University, Columbus, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Medical Center of South Carolina, Charleston, South Carolina

REFERENCES:
- [Background] Diekema DJ, Messer SA, Brueggemann AB, Coffman SL, Doern GV, Herwaldt LA, Pfaller MA. Epidemiology of candidemia: 3-year results from the emerging infections and the epidemiology of Iowa organisms study. J Clin Microbiol. 2002 Apr;40(4):1298-302. doi: 10.1128/JCM.40.4.1298-1302.2002. PMID 11923348
- [Background] Jarvis WR. Epidemiology of nosocomial fungal infections, with emphasis on Candida species. Clin Infect Dis. 1995 Jun;20(6):1526-30. doi: 10.1093/clinids/20.6.1526. PMID 7548503
- [Background] Goodman JL, Winston DJ, Greenfield RA, Chandrasekar PH, Fox B, Kaizer H, Shadduck RK, Shea TC, Stiff P, Friedman DJ, et al. A controlled trial of fluconazole to prevent fungal infections in patients undergoing bone marrow transplantation. N Engl J Med. 1992 Mar 26;326(13):845-51. doi: 10.1056/NEJM199203263261301. PMID 1542320
- [Background] Denning DW. Echinocandins: a new class of antifungal. J Antimicrob Chemother. 2002 Jun;49(6):889-91. doi: 10.1093/jac/dkf045. No abstract available. PMID 12039879
- [Derived] Ostrosky-Zeichner L, Shoham S, Vazquez J, Reboli A, Betts R, Barron MA, Schuster M, Judson MA, Revankar SG, Caeiro JP, Mangino JE, Mushatt D, Bedimo R, Freifeld A, Nguyen MH, Kauffman CA, Dismukes WE, Westfall AO, Deerman JB, Wood C, Sobel JD, Pappas PG. MSG-01: A randomized, double-blind, placebo-controlled trial of caspofungin prophylaxis followed by preemptive therapy for invasive candidiasis in high-risk adults in the critical care setting. Clin Infect Dis. 2014 May;58(9):1219-26. doi: 10.1093/cid/ciu074. Epub 2014 Feb 18. PMID 24550378

RESULTS

PARTICIPANT FLOW:
Groups:
- Prophylaxis: Caspofungin 50 mg IV daily up to 28 days of therapy
- Placebo: Normal Saline 100 cc IV daily
Period: Overall Study
Arm/Group | Prophylaxis | Placebo
Started | 118 | 104
Completed | 117 | 102
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prophylaxis | Placebo | Total
Number analyzed (Participants) | 117 | 102 | 219
Age Continuous [Mean (Standard Deviation); unit: years] | 58.2 (17.5) | 56.7 (16.6) | 57.5 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 41 | 87
  Male | 71 | 61 | 132
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 8 | 15
  Not Hispanic or Latino | 109 | 94 | 203
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 2
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 35 | 35 | 70
  White | 78 | 60 | 138
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 5 | 8
Acute Physiology And Chronic Health Evaluation (APACHE) II score (minimum 0, maximum 71) [Mean (Standard Deviation); unit: Score on a scale] | 25.3 (8.0) | 25.1 (8.7) | 25.2 (8.3)

OUTCOME MEASURES:

1. Primary Outcome: Proven and Probable Invasive Candidiasis Based on Modified Mycoses Study Group/European Organization for Research and Treatment of Cancer (MSG/EORTC) Criteria.
Description: Modified MSG/EORTC criteria for the diagnosis of fungal infections: Proven invasive candidiasis is defined as candidemia, Candida cultured from a sterile site, or histopathological evidence of candida infection. Probable invasive candidiasis is defined as 2 consecutive positive beta glucan levels in the presence of signs and symptoms of infection.
Time Frame: Within 7 days after end of therapy
Population: Modified intent-to-treat population, defined as subjects who received at least one dose of study drug and did not have baseline invasive candidiasis.
Measure: Number; unit: percent of participants
Groups:
- Prophylaxis: Caspofungin 50mg IV daily
Arm/Group | Prophylaxis | Placebo
Number analyzed (Participants) | 102 | 84
percent of participants | 9.8 | 16.6
Statistical Analysis 1: Comparison: Prophylaxis vs Placebo; Test type: Superiority or Other; p = 0.14, Cochran-Mantel-Haenszel; APACHE II Stratified

2. Secondary Outcome: Incidence of Proven Invasive Candidiasis by MSG/ EORTC Criteria.
Time Frame: Within 7 days of end of therapy
Reporting Status: Not Posted

3. Secondary Outcome: All Cause Mortality
Time Frame: Within 7 days of end of therapy
Reporting Status: Not Posted

4. Secondary Outcome: Initiation of Other Antifungals
Time Frame: Within 7 days after end of therapy
Reporting Status: Not Posted

5. Secondary Outcome: Time to Development of Proven or Probable Invasive Candidiasis
Time Frame: Within 7 days after end of therapy
Reporting Status: Not Posted

6. Secondary Outcome: Incidence of Proven and Probable Invasive Fungal Infections Other Than Invasive Candidiasis.
Time Frame: Within 7 days after end of therapy
Reporting Status: Not Posted

7. Secondary Outcome: Time to Beta Glucan Negativity in Pre-emptive Phase.
Time Frame: Within 14 days after end of therapy
Reporting Status: Not Posted

8. Secondary Outcome: Incidence of Complete and Partial Response by Clinical and Microbiological or Serological Evidence for Subjects on the Pre-emptive Therapy Phase.
Time Frame: Within 14 days after end of therapy
Reporting Status: Not Posted

9. Secondary Outcome: Hospital Metrics (to be Evaluated Separately for Prophylaxis and Pre-emptive Therapy Phases); Length of Stay in the Hospital, Length of Stay in the ICU, and the Costs Data for the ICU Stay and the Hospitalization, if Available.
Time Frame: Hospital discharge
Reporting Status: Not Posted

10. Secondary Outcome: Subjects Who Discontinue Study Therapy Due to a Drug-related Adverse Event
Time Frame: Up to 14 days after end of therapy
Population: Safety population, defined as all subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Prophylaxis | Placebo
Number analyzed (Participants) | 117 | 102
participants | 2 | 2

11. Secondary Outcome: Subjects With 1 or More Serious Drug-related Adverse Event(s)
Time Frame: Up to 14 days after end of therapy
Population: Safety population, defined as all subjects who received at least one dose of study drug.
Measure: Number; unit: participants
Arm/Group | Prophylaxis | Placebo
Number analyzed (Participants) | 117 | 102
participants | 1 | 0

ADVERSE EVENTS:
Time Frame: Within 14 days of completion of study therapy.
Arm/Group | Prophylaxis | Placebo
Serious Adverse Events (participants affected / at risk) | 33/117 | 28/102
Other Adverse Events (participants affected / at risk) | 106/117 | 87/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prophylaxis (N=117) | Placebo (N=102)
Atrioventricular extrasystoles (Cardiac disorders) | 1 | 0
Bradyarrhythmia (Congenital, familial and genetic disorders) | 0 | 1
Bradycardia (Cardiac disorders) | 0 | 1
Cardiac arrest (Cardiac disorders) | 3 | 3
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Cardiomyopathy acute (Cardiac disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 4 | 1
Electromechanical dissociation (Cardiac disorders) | 0 | 1
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 2 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Multi-organ failure (General disorders) | 0 | 2
Sudden death (General disorders) | 0 | 1
Abdominal sepsis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 8 | 3
Septic shock (Infections and infestations) | 7 | 0
Transaminases increased (Investigations) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain stem infarction (Nervous system disorders) | 1 | 0
Grand mal convulsion (Nervous system disorders) | 1 | 0
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Haemorrhagic stroke (Nervous system disorders) | 0 | 1
Ischaemic stroke (Nervous system disorders) | 0 | 1
Metabolic encephalopathy (Nervous system disorders) | 1 | 0
Spinal cord infarction (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Deep vein thrombosis (Vascular disorders) | 1 | 0
Flushing (Vascular disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1
Shock (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Prophylaxis (N=117) | Placebo (N=102)
Anaemia (Blood and lymphatic system disorders) | 14 | 13
Leukocytosis (Blood and lymphatic system disorders) | 14 | 7
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 4
Diarrhoea (Gastrointestinal disorders) | 6 | 6
Pyrexia (General disorders) | 18 | 6
Bacteraemia (Infections and infestations) | 5 | 7
Sepsis (Infections and infestations) | 9 | 5
Septic shock (Infections and infestations) | 8 | 0
Blood urea increased (Investigations) | 6 | 3
Hepatic enzyme increased (Investigations) | 13 | 3
Hyperglycaemia (Musculoskeletal and connective tissue disorders) | 6 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 3 | 6
Hypoglycaemia (Metabolism and nutrition disorders) | 9 | 7
Hypokalaemia (Metabolism and nutrition disorders) | 11 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 4 | 6
Hypophosphataemia (Metabolism and nutrition disorders) | 8 | 3
Agitation (Psychiatric disorders) | 7 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 11 | 4
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 7 | 3
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 | 4
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3 | 6
Deep vein thrombosis (Vascular disorders) | 10 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less